CLINICAL TRIAL: NCT00418184
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Study of The Efficacy and Safety of Phosphatidylserine-Omega3 in Children With Attention-Deficit/ Hyperactivity Disorder
Brief Title: The Efficacy and Safety of Phosphatidylserine-Omega3 in Children With Attention-Deficit/ Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enzymotec (Industry)
Responsible Party: Manor Yonatan, Enzymotec LTD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS-Omega3-2
Record Dates: First submitted 2006-12-31; First posted 2007-01-04 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD; inattentive; impulsive; hyperactive; poor academic performance; poor self-discipline; low self-esteem
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Phosphatidylserine-Omega3
- 2 (Placebo Comparator)
  Interventions: Other: Colored cellulose tainted with fishy odor

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine-Omega3 — Phosphatidylserine-Omega3 conjugate capsules. Weeks 0-15: 300 mg/day. weeks 16-30: 150 mg/day and a 150 mg/day one year follow-up.
  Arms: 1
Other: Colored cellulose tainted with fishy odor — as arm 1
  Arms: 2

SUMMARY:
The primary objective of this trial is to determine whether an oral administration of Phosphatidylserine-Omega3 would significantly improve the clinical symptoms of children suffering from ADHD. Both the behavior and the academic achievements aspects will be evaluated. In addition, we intend to measure side-effects and adverse events and to examine the possible correlation between biochemical and behavioral alterations.

DETAILED DESCRIPTION:
This study is a single-center, double-blind, randomized, placebo-controlled 15-weeks duration trial to assess safety and efficacy of Phosphatidylserine-Omega3 in children diagnosed with ADHD, according to the DSM-IV. Following screening, the subjects will be randomized to one of two treatment groups:Phosphatidylserine-Omega3 or placebo, in a 2:1 manner. This will be followed by an open-label extension, in which Phosphatidylserine-Omega3 will be administered to all eligible participants.

Primary measures of attention and behavior will be evaluated using Conners Rating Scale (CRS) teacher- rating scales. As a secondary endpoint, the attention and behavior will be measured by CRS and strength and difficulties questionnaires (SDQ) parental- and SDQ teacher-rating scales, assessment a continuous performance test (TOVA), and parental Child Health questionnaire (CHQ). Improvement in ADHD symptoms will be evaluated by Clinical Global of Impression - Improvement (CGI-I). Finally, tolerability will be monitored using Barkley Side Effects Rating Scale (SERS) and biochemical parameters, such as fatty acid profile and monoamines metabolites will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Parental written informed consent.
2. Having a teacher that is familiar with the child and parent and willing to participate.
3. Age: 13≥ years ≥6
4. Gender: male and female
5. Diagnosis: ADHD diagnosed by:

   Teacher-rated Attention-Deficit/ Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) School Version at least 1.5 standard deviations (SD) above the norm for the patient's age and gender, Confirmed assessment by Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL),
6. Clinical Global Impression of Severity of illness (CGI-S) rating of 4 or higher (moderately ill or worse),
7. Language: Subjects, parents, and teachers must be able to read, write and speak Hebrew
8. Normal weight and height according to the Israeli standards
9. Attending full-time to school.

Exclusion Criteria:

1. Females who had reached menarche and presented three regular menstrual cycles; the definition of regular menstrual cycles: an average length of the cycle between 22 and 41 days, either none or a single cycle with a length less than 22 or more than 41 days during the past year
2. History or current diagnosis of any serious systemic (e.g., diabetes, hyper/hypothyroidism, etc.) or neurological condition (e.g., epilepsy, brain tumors, etc.)
3. Failed to respond to 2 or more adequate courses (dose and duration) of stimulant therapy for ADHD
4. Pervasive developmental disorder or Non-verbal Learning Disability
5. Schizophrenia, or other psychotic disorders (DSM-IV axis I)
6. Any evidence of suicidal risk, any current psychiatric comorbidity that required psychiatric pharmacotherapy
7. History of alcohol or substance abuse as defined by DSM-IV criteria
8. Consumption of >250 mg/day of caffeine
9. Blindness
10. History of allergic reactions or sensitivity to marine products (fish and seafood), soy or corn as well as any illness which may jeopardize the participants health or limit their successful trial completion.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Weizman, MD, Study Director — Head of the Research Department, Geha Mental Health Center, Rabin Medical Center
Locations (1):
- ADHD Unit, Petach-Tiqva, Israel

REFERENCES:
- [Derived] Manor I, Magen A, Keidar D, Rosen S, Tasker H, Cohen T, Richter Y, Zaaroor-Regev D, Manor Y, Weizman A. The effect of phosphatidylserine containing Omega3 fatty-acids on attention-deficit hyperactivity disorder symptoms in children: a double-blind placebo-controlled trial, followed by an open-label extension. Eur Psychiatry. 2012 Jul;27(5):335-42. doi: 10.1016/j.eurpsy.2011.05.004. Epub 2011 Jul 31. PMID 21807480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children at the age of 6-13 years were screened at the "Geha mental health center", Israel, for participation in the study. Recruitment of participants was achieved by vast advertisement in newspapers, internet and in practitioners clinics. Participants enrollment period March 2007 to March 2008
Groups:
- PS Omega 3 Conjugate: The daily dosage consisted of 4 capsules of PS-Omega3, providing 300 mg Phosphatidylserine per day.
- Placebo: Double-blind: Cellulose (4 capsules per day). Open-label: PS-omega3
Period: Double-blind Phase
Arm/Group | PS Omega 3 Conjugate | Placebo
Started | 137 | 63
Completed | 110 | 52
Not Completed | 27 | 11
Not completed — Withdrawal by Subject | 22 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Poor compliance | 3 | 1
Period: Open-label Phase
Arm/Group | PS Omega 3 Conjugate | Placebo
Started | 102 (3 were not included due to low compliance in the double blind phase, 5 didn't want to participate.) | 48 (1 was not included due to low compliance in the double blind phase, 3 didn't want to participate.)
Completed | 97 (5 dropped out) | 43 (5 dropped out)
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PS Omega 3 Conjugate | Placebo | Total
Number analyzed (Participants) | 137 | 63 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.10 (1.89) | 9.24 (1.77) | 9.15 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 22 | 67
  Male | 92 | 41 | 133
Clinical Global Impression of Severity (CGI-S) [Number; unit: Participants] — The CGI is an observer-rated scale that measures illness severity.The clinician evaluates the patient relative to his past experience with other patients with the same diagnosis.The ratings of CGI-S are: 1 = not ill at all, 2 = a borderline case, 3 = only mildly ill, 4 = moderately ill, 5 = seriously ill and 6 = extremely seriously ill.
  Participants
    Moderately ill (score 4) | 83 | 36 | 119
    Seriously ill (score 5) | 50 | 27 | 77
    Extremely seriously ill (score 6) | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Conners Rating Scale - School Version
Description: A questionnaire that assesses symptoms of ADHD in children and adolescents according to the DSM-IV guidelines. It consists of questions on classroom behavior. Based on the questionnaire results, subscales and global indexes are calculated, including restless-impulsive index, emotional lability index and hyperactive/impulsive subscale. The lowest scale score is 40 (best)and the highest is 90 (worse). Usually, a score below 62 is considered normal and a score above 62 is considered abnormal.
Time Frame: change from baseline in conners raiting scale at 15 weeks
Population: The analysis includes per-protocol (PP) population. Out of the 162 children who completed the study, 15 children were excluded from PP analysis due to low compliance or protocol violation.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | PS Omega 3 Conjugate | Placebo
Number analyzed (Participants) | 100 | 47
Scores on a scale
  Conners Global Index: restless impulsivity | -0.44 (1.04) | -1.73 (1.67)
  Conners Global index: Emotional Lability | -2.63 (1.18) | -0.63 (1.77)
  Hyperactivity-impulsivity | -0.62 (1.09) | -0.46 (1.25)

2. Secondary Outcome: Conners Rating Scale - Home Version
Description: A questionnaire that assesses symptoms of ADHD in children and adolescents according to the DSM-IV guidelines. It consists of questions on the childs home behavior. Based on the questionnaire results, subscales and global indexes are calculated, including restless-impulsive index, emotional lability index and hyperactive/impulsive subscale. The lowest scale score is 40 (best)and the highest is 90 (worse). Usually, a score below 62 is considered normal and a score above 62 is considered abnormal.
Time Frame: change from baseline in conners raiting scale at 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | PS Omega 3 Conjugate | Placebo
Number analyzed (Participants) | 100 | 47
Scores on a scale
  Conner's Global restless-impulsivity | -5.19 (1.00) | -1.71 (1.72)
  Conner's Global Index:Emotional lability | -3.54 (1.08) | -5.56 (1.80)
  DSM-IV: Hperactivity impulsivity | -4.23 (1.15) | -2.62 (1.77)

3. Secondary Outcome: Strength and Difficulties Questionnaires - School Version
Time Frame: on weeks 0,15
Reporting Status: Not Posted

4. Secondary Outcome: Strength and Difficulties Questionnaires - Home Version
Time Frame: on weeks 0,15
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Global Impression of Improvement
Time Frame: on weeks 0,15
Reporting Status: Not Posted

6. Secondary Outcome: Test of Variables of Attention (TOVA)
Time Frame: on weeks 0,15
Reporting Status: Not Posted

7. Secondary Outcome: Child Health Questionnaire (CHQ)- Parent-completed Form 50
Time Frame: on weeks 0,15
Reporting Status: Not Posted

8. Secondary Outcome: Plasma and Red Blood Cells Fatty Acid Profile
Time Frame: on weeks 0,15
Reporting Status: Not Posted

9. Secondary Outcome: Blood Monoamines Metabolism
Time Frame: on week 0, 15
Reporting Status: Not Posted

10. Secondary Outcome: Vital Signs
Time Frame: on weeks 0,15
Reporting Status: Not Posted

11. Secondary Outcome: Essential Fatty Acid (EFA)-Deficiency Symptoms
Time Frame: on weeks 0,15
Reporting Status: Not Posted

12. Secondary Outcome: Barkley Side Effects Rating Scale (SERS)
Time Frame: on weeks 0,15
Reporting Status: Not Posted

13. Secondary Outcome: Complete Blood Counts
Time Frame: on weeks 0,15
Reporting Status: Not Posted

14. Secondary Outcome: Biochemical Parameters in Blood - Liver Functions (SGPT, SGOT, Total Bilirubin), Kidney Functions (BUN, Creatinine), Na, K, Cl, Ca
Time Frame: on weeks 0,15
Reporting Status: Not Posted

15. Secondary Outcome: Lipid Profile (Cholesterol, HDL, Triglycerides)
Time Frame: on weeks 0,15
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PS Omega 3 Conjugate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/63
Other Adverse Events (participants affected / at risk) | 6/137 | 1/63
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS Omega 3 Conjugate (N=137) | Placebo (N=63)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other